CLINICAL TRIAL: NCT05632822
Title: Predictive Value of Diaphragm Function Monitoring for Weaning in Mechanically Ventilated Patients: a Prospective Observational Cohort Study
Brief Title: Value of Diaphragm Function Predicting Weaning From Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K2603
Record Dates: First submitted 2022-11-08; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Weaning Failure; Diaphragm Defect
Keywords: Weaning Failure; Diaphragm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SBT failure: The SBT was considered to be a failure if at least one the following criteria was present: (1) blood oxygen saturation (SpO2) of <90 % with a fraction of inspired oxygen (FiO2) of≥50 %; (2) acute respiratory distress (RR≥40/min, agitation, cyanosis); (3) systolic arterial blood pressure of ≥180 mmHg; (4) cardiac arrhythmias; (5) respiratory acidosis [pH<7.32 with an arterial carbon dioxide tension (PaCO2) of ≥50 mmHg].
- SBT success: If none of these failure criteria was present, the SBT was considered as successfully completed.

SUMMARY:
The reason of failure of weaning from mechanical ventilation is that their respiratory loads exceeding the capacity of their respiratory muscles. The electric activity of diaphragm (EADI) allows quantification of the neural respiratory drive to the diaphragm. The aim of this study is to evaluate diaphragmatic ultrasound related parameters and electric activity of diaphragm (EADI) during SBT and postural changes to predict weaning outcome.

DETAILED DESCRIPTION:
The reason of failure of weaning from mechanical ventilation is that their respiratory loads exceeding the capacity of their respiratory muscles. The aim of this study is to evaluate diaphragmatic ultrasound related parameters and electric activity of diaphragm (EADI) during SBT and postural changes to predict weaning outcome. EADI catheter consists of a nasogastric feeding tube equipped with a multiple-array esophageal electrode that provides real time access to EADI.

Patients intubated and ventilated for at least 48 h were eligible for inclusion in the study.

After the ward physician judged that the patients' condition met the offline standard, patients were prepared to conduct spontaneous breathing trial (SBT). All recruited patients were placed EADI catheter.

The protocol started with patients ventilated on a PSV of 10 cm H2O above a positive end-expiratory pressure (PEEP) of 4-5 cm H2O. Then record ventilator parameters, EADI parameters (including maximum EADI, minimum EADI, area under the curve of the EADI during inspiratory time) and diaphragmatic ultrasound related parameters (diaphragm thickness and diaphragm displacement) respectively in the semi-seated and supine positions. Then assist was removed and a 30-minute SBT was performed with continuous positive airway pressure (CPAP) of 4-5 cm H2O at the previous level of FiO2. At 0, 1, 5, 10, 20 and 30 minutes into the SBT vital signs, ventilatory parameters (including RR, Vt, Ppeak, PEEP, P0.1, MV) were collected. Arterial blood gases were sampled at the start and the end of the SBT.

The SBT was considered to be a failure if at least one the following criteria was present: (1) blood oxygen saturation (SpO2) of <90 % with a fraction of inspired oxygen (FiO2) of≥50 %; (2) acute respiratory distress (RR≥40/min, agitation, cyanosis); (3) systolic arterial blood pressure of ≥180 mmHg; (4) cardiac arrhythmias; (5) respiratory acidosis [pH<7.32 with an arterial carbon dioxide tension (PaCO2) of ≥50 mmHg]. If none of these failure criteria was present, the SBT was considered as successfully completed.

Patient was reconnected if signs of intolerance were present. The separation from the ventilator and the endotracheal tube was considered a success when spontaneous breathing could be sustained without any form of ventilatory support at 48h after extubation. Failure cases included patients who failed the SBT and patients requiring reintubation or any form of ventilator support (including non-invasive ventilation for post-extubation acute respiratory failure) during the first 48 h after extubation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old Patients with acute respiratory failure and endotracheal intubation Invasive ventilator time ≥48 hours Switched to auxiliary ventilation mode and have weaning plan.

Exclusion Criteria:

Patients with severe neuromuscular diseases Patients treated with muscle relaxants Patients who have been or are about to be discontinued from life support Patients with esophageal and fundus varicose veins, digestive tract perforation or gastric tube insertion after upper digestive tract surgery contraindicated Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were intubated and ventilated for at least 48 h, who need to conduct weaning protocol.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
EADI ( diaphragm electrical activity) | 30 minutes since SBT was conducted
  Utilizing NAVA catheter, the EADI allows quantification of the neural respiratory drive to the diaphragm.

SECONDARY OUTCOMES:
Diaphragm Neurodisplacement Efficiency | 30 minutes since SBT was conducted
  Diaphragm Neurodisplacement Efficiency (NDE) is the ratio between diaphragm displacement and EAdi. It is uesd to describe the efficiency of EADI transferred to diaphragm displacement.
Neuroventilatory Efficiency | 30 minutes since SBT was conducted
  Neuroventilatory Efficiency is the ratio of tidal volume and diaphragm electrical activity (Vt/EAdi) .

CONTACTS AND LOCATIONS:
Overall Officials: Li Weng, Dr, Study Director — Director of department
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diao S, Li S, Dong R, Jiang W, Wang C, Chen Y, Wang J, He S, Wang Y, Du B, Weng L. The diaphragmatic electrical activity during spontaneous breathing trial in patients with mechanical ventilation: physiological description and potential clinical utility. BMC Pulm Med. 2024 May 30;24(1):263. doi: 10.1186/s12890-024-03077-8. PMID 38816810